CLINICAL TRIAL: NCT03277287
Title: Assessment of Fractional CO2 Laser in Treatment of Post-surgical Scarring of Cleft Lip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Shadad Rateb Mohamed, Resident doctor, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CO2 laser in cleft lip scar
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Cleft Lip Post-surgical Scar

STUDY DESIGN:
Intervention Model Description: Prospective comparative study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Fractional CO2 laser will be applied on cleft lip scar 3 weeks post-surgical
  Interventions: Radiation: Fractional CO2 laser
- Group B (Experimental): Fractional CO2 laser will be applied on cleft lip scar 3 months post-surgical
  Interventions: Radiation: Fractional CO2 laser
- Group C (No Intervention): No intervention

INTERVENTIONS:
Radiation: Fractional CO2 laser — Fractional CO2 laser will be applied in cleft lip scar to assess and evaluate the later appearance of the scar
  Arms: Group A; Group B

SUMMARY:
This is a prospective comparative study on 120 patients divided to three groups. Group A: 40 patients laser will be applied 3 weeks post-surgical. Group B: 40 patients laser will be applied 3 months post surgical. Group C: 40 patients as a control not treated with laser from 2017 to 2020 which will be conducted on patients with post-surgical cleft lip repair scaring.

All patients will have 5-7 sessions with 4 weeks interval.

Photographic documentation and evaluation of the scar will occur every 4 weeks.

DETAILED DESCRIPTION:
The carbon dioxide laser (CO2 Laser) was one of the earliest gas lasers to be developed. It was invented by Kumar Patel of Bell Labs in 1964.

CO2 laser is the highest power continuous wave lasers that are currently available which produces a beam of infrared light with the principal wavelength bands centering on 9.4 and 10.6 micrometers. Patel, C. K. N. (1964).

When CO2 beam of light is selectively applied to the skin, it heats and vaporizes various layers of skin, instantly treating damaged skin and wrinkles while smoothing out the surface of the skin.

The skin remodeling occurs with new skin and collagen growth. The healing typically involves an open surface which takes weeks to heal and typically results in loss of the baseline pigmentation leading to variable lightening of skin. Dover, J. S. (2012) Fractional CO2 laser resurfacing is a revolutionary delivery system that provides dramatic skin improvement without surgery. Matrix combines the benefits of CO2 laser by using micro laser columns "points of light" to treat the epidermis and dermal layers of your skin.

Bernstein et al, (1997) Cleft lip is a form of lip malformation that occurs very early in pregnancy, the incidence of cleft lip in the population is approximately 0.5-2 in 1000 live births. Male children are affected more often than female children.

Michalski AM et al, (2015). Because each cleft is unique, definitive repair of the cleft lip should be individualized as Mirault, Le Mesurier, Tennison, and Millard.

Stal S et al, (2009)

ELIGIBILITY:
Inclusion Criteria:

* Any age with acceptable scar which would not need further revision.
* Group A: three weeks after repair & group B: three months after repair with no hypertrophy, erythema or any other scar complication.

Exclusion Criteria:

* Any case with deformity needing further surgical interference.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Vancouver scar scale | 5 -7 months
  It assess four variables:vascularity , height/thickness , pigmentation , pliability

SECONDARY OUTCOMES:
Visual analogue scale | 5-7 months
  This depends on 5 independent medical and nonmedical personnel rating results on a graded scale 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Wagdi Ali, Dr, Study Director — Assiut University; Mohamed Elshazly, Prof., Principal Investigator — Assiut University
Locations (1):
- Mohamed shadad, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shadad M, Ali WM, Fayyaz GQ, El-Shazly M. Use of Fractional CO2 Laser in Cleft Lip Scars: Does It Make a Difference? Ann Plast Surg. 2021 May 1;86(5):536-539. doi: 10.1097/SAP.0000000000002511. PMID 32826442